CLINICAL TRIAL: NCT06160050
Title: Randomized Control Trial of the Breakthrough Parenting Curriculum: Transforming Trauma Across Generations
Brief Title: PRESERVE & CONNECT: Impact Study of the BPC
Acronym: (BPC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Jessica Strolin-Goltzman, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2648
Record Dates: First submitted 2023-06-23; First posted 2023-12-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Child Maltreatment; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The Preserve and Connect Project will be a two arm (BPC+ TAU vs TAU) parallel randomized clinical trial to determine the efficacy of the BPC and establish the evidence base to allow the BPC to be listed on the Title IV-E Clearing House. Participants will be recruited from individuals seeking treatment from our community partners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPC (Experimental)
  Interventions: Behavioral: Breakthrough Parenting Curriculum: Transforming trauma across generations
- Treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Breakthrough Parenting Curriculum: Transforming trauma across generations — The BPC (Breakthrough Parent Curriculum): Navigating Trauma Across Generations is a 10 module course adapted from the NCTSN training called Caring for Children Who Have Experienced Trauma: A Workshop for Resource Parents (RPC). The BPC is specifically designed for parents who have been involved with (or are at risk for being involved with)the child welfare system. The course provides information about the impact of trauma on the development, attachment, emotions and behaviors of children while holding space for parents to learn together about concrete strategies for managing daily and ongoing challenges and enhancing their relationships with their children. All while acknowledging the challenges of parenting a child who has experienced trauma, while having experienced your own trauma.
  Arms: BPC

SUMMARY:
The PRESERVE & CONNECT project is a multi-site randomized control trial of the Breakthrough Parenting Curriculum: Navigating Trauma Across Generations (BPC) in rural and racially and ethnically diverse communities in Vermont and Connecticut.

DETAILED DESCRIPTION:
The proposed study will determine the efficacy of the BPC at improving the lives of families with a significant history of trauma and establish the evidence base to allow the BPC to be listed on the Title IV-E Clearing House. The specific research questions that will be answered as are as follows:

Question 1: Does the BPC improve Child Safety? Hypothesis 1a: Parents who complete the BPC will have fewer substantiated of child maltreatment as per administrative records.

Hypothesis 1b: Parents who complete the BPC will report less psychologically aggressive and abusive parenting behaviors (Parenting Scale).

Question 2: Does the BPC improve Child Permanency? Hypothesis 2a: Parents who complete the BPC will have fewer out of family placements and placement disruptions as per administrative records.

Hypothesis 2b: Parents who complete the BPC will have stability or permanency with their family of origin as per administrative records.

Question 3: Does the BPC improve Child Well-Being? Hypothesis 3: Parents who complete the BPC will report improved behavioral and emotional functioning of their children (Strength and Difficulties Questionnaire).

Question 4: Does the BPC improve Adult Well-Being? Hypothesis 4a: Parents who complete the BPC will report improved use of parenting practices to improve the functional relationship with their children (Parenting Self-Efficacy Scale; Parent Stress Index, Parent-Child Relationship Scales).

Hypothesis 4b: Parents who complete the BPC will report improved understanding of the influence of trauma on their parenting behaviors and wellness (Trauma-Informed Knowledge and Parenting Skills Survey).

Question 5: Are the improvements of the BPC associated with demographic factors? Exploratory Analysis 5a: Examine the association between measures of child safety, child well-being, child permanency, and adult well-being and measures of acculturation.

Exploratory Analysis 5a: Examine the association between measures of child safety, child well-being, child permanency, and adult well-being and measures of acculturation

ELIGIBILITY:
Inclusion Criteria:

- Parents involved in, or at risk of involvement in, the child welfare system.

Exclusion Criteria:

* active psychosis without medication stabilization
* ongoing major depressive episodes
* active suicidal ideation
* active homicidal ideation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Child Safety | up to 6 months
  substantiated reports of child maltreatment as per administrative records
Child Permanency | up to 6 months
  out of family placements and placement disruptions as per administrative records. Total amount of each type of placement.
Child Well-being | 10 weeks
  behavioral and emotional functioning of their children (Strength and Difficulties Questionnaire).
Parenting Self-Efficacy Scale | 10 weeks
  Scores range from 0-160. Higher scores indicate more self efficacy

SECONDARY OUTCOMES:
Parental Stress Index | 10 weeks
  Parent Stress Index Self-Report Measure
Trauma-Informed Knowledge and Parenting Skills Survey | 10 weeks
  understanding of the influence of trauma on their parenting behaviors and wellness

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Connecticut, Hartford, Connecticut
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided